CLINICAL TRIAL: NCT06827990
Title: Evaluation of the GORE® Ascending Stent Graft in the Treatment of De Novo Type A Aortic Dissections
Brief Title: GORE® Ascending Stent Graft in the Treatment of De Novo Type A Aortic Dissections
Acronym: ARISE III
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASG 24-02
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Primary (Experimental): A hypothesis driven analysis of the safety and effectiveness of the GORE® Ascending Stent Graft (ASG) device alone in the ascending aorta. Dissection chronicity in the primary arm must be 30 days or less from symptom onset to index endovascular procedure.
  Interventions: Device: GORE® Ascending Stent Graft (ASG device)
- Secondary (Experimental): Descriptive analysis of use of the ASG device in patients who are not eligible for treatment in the primary arm. Dissection chronicity up to 90 days from symptom onset until the first study procedure is allowed in the secondary arm.
  Interventions: Device: GORE® Ascending Stent Graft (ASG device)

INTERVENTIONS:
Device: GORE® Ascending Stent Graft (ASG device) — Endovascular aortic repair of the ascending aorta

SUMMARY:
To assess the safety and effectiveness of the ASG device in the treatment of de novo Type A aortic dissections.

DETAILED DESCRIPTION:
This pivotal investigation is a prospective, multicenter, non-randomized, single-arm study to evaluate the safety and effectiveness of the ASG device for the treatment of de novo Type A aortic dissections in patients considered to be high-risk for open surgical repair.

ELIGIBILITY:
Inclusion Criteria - Primary Arm:

The subject is/has:

1. De novo Type A aortic dissection (≤30 days from symptom onset to index endovascular procedure) compatible with the treatment requirements of the ASG device.
2. Primarily intended to be treated by placement of the ASG device in the ascending aorta. Distal adjunctive procedures not in contact with the ASG device may be performed during the index endovascular procedure at the discretion of the Investigator.
3. Anatomic compatibility of the ascending aorta required for implanting the ASG device:

   a) Proximal Aortic Landing Zone: i. Primary entry tear must be in the ascending aorta and ≥ 2 cm distal to the most distal coronary artery ostium.

   ii. Total aortic diameter between 27mm - 48mm iii. Landing zone cannot be heavily calcified or thrombosed. b) Distal Aortic Landing Zone: i. Primary entry tear must be in the ascending aorta and ≥ 2 cm proximal to BCA ostium.

   c) Adequate aortic length
4. The Aortic Treatment Team (as defined by the protocol) attest endovascular repair is in the best interest of the patient AND considers the patient to be high-risk for open surgical repair by meeting at least one of the following criteria:

   1. ≥80 years of age
   2. Body mass index (BMI) ≥ 35 kg/m2
   3. History of Respiratory Insufficiency (defined by home O2 usage, exertional dyspnea, imaging evidence of COPD, previous evidence of compromised pulmonary function tests (PFT) on spirometry or other factors as determined by the Investigator)
   4. Prior Cardiac Surgery
   5. Hostile Chest (VARC-2 Definition)
   6. Clinical Frailty Scale 3-7
   7. Clinical malperfusion (head, gut, lower extremity)
   8. Transfusion is not possible (e.g., Jehovah's Witness)
   9. Renal Dialysis prior to aortic dissection
   10. Chronic renal insufficiency (eGFR<60 without dialysis or other documented history of chronic kidney disease prior to dissection)
5. Age ≥18 years at time of informed consent signature.
6. Adequate vascular access via transfemoral or retroperitoneal approach.
7. Informed Consent Form (ICF) signed by the subject or legally authorized representative.
8. Agrees to comply with protocol requirements, including imaging and 5-year follow-up, as the subject's condition allows.

Exclusion Criteria - Primary Arm

The subject is/has:

1. Mechanical heart valve in the aortic position.
2. Aortic insufficiency grade 3 or greater confirmed during TEE pre-implant.
3. Indwelling intravascular device that would interfere with or result in contact with planned repair (e.g., contiguous arch graft, LVAD, TAVR device in continuity with aortic tear).
4. Known degenerative connective tissue disease (e.g., Marfan's or Ehler-Danlos Syndrome).
5. Participation in investigational drug or medical device study within one year of enrollment unless approved by the Sponsor.
6. Known history of drug abuse within one year of treatment which would affect the ability to obtain follow-up.
7. Pregnant at time of procedure.
8. Active infected aorta, mycotic aneurysm.
9. Active systemic infection (e.g., infection requiring treatment with parenteral anti-infective medication).
10. Life expectancy <12 months due to presence of another comorbid condition.
11. Known sensitivities or allergies to the device materials (Previous instance of Heparin Induced Thrombocytopenia type 2 [HIT-2], known hypersensitivity to heparin, or a history of a hypercoagulability disorder and/or state should be considered exclusion if treatment plan includes implant of a TBE device).
12. Known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment.
13. Coronary malperfusion.
14. Catastrophic neurological complications in the 30 days prior to the dissection diagnosis (e.g., progressively worsening symptoms, coma, Glasgow Coma Scale <=8).
15. Aortic fistula.
16. In circulatory shock (e.g., systolic blood pressure <80 mmHg without inotropes, base deficit > -10 mmol/L or -10 mEq/L) at any time prior to the initiation of the index endovascular procedure.
17. In extreme hemodynamic compromise requiring cardiopulmonary resuscitation at any time prior to the initiation of the index endovascular procedure.
18. Clinical or radiographic signs of bowel infarction, gastrointestinal hemorrhage, or bowel necrosis (as determined by the implanting physician based on imaging observations, peritoneal signs, surgical exploration, elevated serum lactate levels, low pH, and/or acidosis) at any time prior to the initiation of the index endovascular procedure.

Inclusion Criteria - Secondary Arm

The subject is/has:

1. De novo Type A aortic dissection (≤90 days from symptom onset until first study procedure) compatible with the treatment requirements of the ASG device alone or the ASG device in combination with the TBE device in the Zone 0 position.
2. Primarily intended to be treated by placement of the ASG device in the ascending aorta or ASG device in combination with the TBE device in the ascending aorta and aortic arch. Distal adjunctive procedures not in contact with the ASG device may be performed during the index endovascular procedure at the discretion of the Investigator.
3. Anatomic requirements for intended treatment with the ASG device alone or in combination with the TBE device.

   a) Anatomic compatibility required for implanting the ASG device (Intended treatment with ASG device alone) i. Proximal Aortic Landing Zone:
   1. Primary entry tear must be in the ascending aorta and ≥ 2 cm distal to the most distal coronary artery ostium.
   2. Total aortic diameter between 27mm - 48mm.
   3. Landing zone cannot be heavily calcified or thrombosed. ii. Distal Aortic Landing Zone:

   <!-- -->

   1. Primary entry tear must be in the ascending aorta and ≥ 2 cm proximal to BCA ostium.

      iii. Adequate aortic length
   2. Anatomic compatibility required for implanting the ASG device (Intended treatment with ASG device and TBE device) i. Proximal Aortic Landing Zone:

   <!-- -->

   1. Primary entry tear must be identified in Zone 0-5.
   2. Landing zone is native aorta.
   3. Primary entry tear location is ≥2cm distal to the most distal coronary artery ostium.
   4. Proximal landing zone must be ≥2cm in the ascending aorta.
   5. Landing zone cannot be heavily calcified or thrombosed.
   6. Total aortic landing zone diameter 27mm - 48mm. ii. Branch Vessel Landing Zone:

   <!-- -->

   1. Length of ≥2.5 cm proximal to first major branch vessel.
   2. Target branch vessel inner diameters of 11-18 mm.
   3. Target branch vessel landing zone must be in native vessel that cannot be heavily calcified or thrombosed.
   4. The distal 15mm landing zone cannot be dissected.
4. The Aortic Treatment Team (as defined by the protocol) attest endovascular repair is in the best interest of the patient AND considers the patient to be high-risk for open surgical repair by meeting at least one of the following criteria:

   1. ≥80 years of age
   2. BMI ≥ 35 kg/m2
   3. History of Respiratory Insufficiency (defined by home O2 usage, exertional dyspnea, imaging evidence of COPD, previous evidence of compromised PFTs on spirometry or other factors as determined by the Investigator)
   4. Prior Cardiac Surgery
   5. Hostile Chest (VARC-2 Definition)
   6. Clinical Frailty Scale 3-9
   7. Clinical malperfusion (head, gut, lower extremity)
   8. Transfusion is not possible (e.g., Jehovah's Witness)
   9. Renal Dialysis prior to aortic dissection
   10. Chronic renal insufficiency (eGFR<60 without dialysis or other documented history of chronic kidney disease prior to dissection)
5. Age ≥18 years at time of informed consent signature.
6. Adequate vascular access via transfemoral or retroperitoneal approach.
7. Informed Consent Form (ICF) signed by the subject or legally authorized representative.
8. Agrees to comply with protocol requirements, including imaging and 5-year follow-up, as the subject's condition allows.

Exclusion Criteria - Secondary Arm:

The subject is/has:

1. Mechanical heart valve in the aortic position.
2. Pregnant at time of procedure.
3. Active infected aorta, mycotic aneurysm.
4. Active systemic infection (e.g., infection requiring treatment with parenteral anti-infective medication).
5. Known sensitivities or allergies to the device materials (Previous instance of Heparin Induced Thrombocytopenia type 2 [HIT-2], known hypersensitivity to heparin, or a history of a hypercoagulability disorder and/or state should be considered exclusion if treatment plan includes implant of a TBE device).
6. Known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 30 Days
  Composite of the following events:
  Death ≤30 days of the index endovascular procedure, or during initial hospitalization, whichever is later
  Disabling Stroke ≤30 days following the index endovascular procedure
Primary Effectiveness Endpoint | 30 Days
  Clinical Success, a composite of:
  Assisted Technical Success (at end of index endovascular procedure)
  Absence of the following (cumulative through 30-days, except as specified):
  Aortic rupture
  Death ≤30days of the index endovascular procedure, or during initial hospitalization, whichever is later
  Study Device Reintervention
  Conversion to open surgical repair

SECONDARY OUTCOMES:
Secondary Endpoint | 1 Year
  Procedural Success
  Treatment Success
  Primary Technical Success (Unassisted)
  SF-36® Physical Component Summary measured at one year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Eric Roselli, MD, Principal Investigator — The Cleveland Clinic
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida, Gainesville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Methodist Hospital Houston, Houston, Texas
  - Baylor Research Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.